CLINICAL TRIAL: NCT01337882
Title: Inhalation of Dilute Biodiesel Exhaust: Acute Vascular and Endothelial Responses
Brief Title: Biodiesel Exhaust, Acute Vascular and Endothelial Responses
Acronym: BEAVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Umeå University (Other)
Responsible Party: Principal Investigator, Jeremy Langrish, Clinical Lecturer and Specialty Registrar in Cardiology, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BEAVER
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Air Pollution; Diesel exhaust; Biodiesel exhaust; Vascular function; Fibrinolysis; Acute vascular and endothelial responses

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diesel exhaust exposure (Experimental): 1 hour exposure to dilute diesel exhaust (approximate PM10 concentration 300 mcg/m3) during intermittent exercise
  Interventions: Other: Forearm venous occlusion plethysmography study
- Biodiesel exhaust exposure (Experimental): 1 hour exposure to dilute biodiesel exhaust (approximate PM10 concentration 300 mcg/m3) during intermittent exercise
  Interventions: Other: Forearm venous occlusion plethysmography study

INTERVENTIONS:
Other: Forearm venous occlusion plethysmography study — Forearm venous occlusion plethysmography to measure forearm blood flow during unilateral intrabrachial infusion of endothelium-dependent (bradykinin [100, 300 & 1000 pmol/min]; acetylcholine [5, 10 & 20 µg/min]) and -independent [sodium nitroprusside [2, 4 & 8 µg/min]; verapamil [10, 30 & 100 µg/min]) vasodilators. Each drug to be infused for 6 mins at each dose in increasing concentrations. 0.9% sodium chloride will be infused for 20 min between each individual drug to allow washout.

SUMMARY:
Exposure to particulate air pollution has been shown to increase cardiovascular mortality and morbidity, and in previous controlled exposure studies has been shown to have acute cardiovascular and respiratory effects. The last decade has seen an unprecedented drive towards finding a bioeconomical and renewable source of fuel in order to reduce our dependence on fossil fuels. Although both biodiesel and bioethanol have emerged as contenders for future fuels, biodiesel remains as the strongest contender within European markets. In 2007 researchers at the EPA released a commentary, which concluded that the assumed correlation between the chemical composition of biodiesel exhaust and a reduction in health effects was only hypothetical. They suggested that there was a clear need for the study of health effects in humans regarding biofuel exhaust. In this project the investigators aim to investigate the cardiovascular, respiratory and inflammatory responses to biofuel exhaust exposure in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 20 healthy, non-smoking subjects, age 20-55 year old, both genders.

All subjects undergo a general health examination and are required to have:

Normal clinical examination Normal EKG Normal routine blood tests Normal lung function

Exclusion Criteria:

* Cardiovascular disease
* Diabetes Mellitus
* Asthma and/or allergy
* Respiratory infection within 3 weeks of the study
* Antioxidant- and/or vitamin supplementation within 2 weeks prior to, as well as during the course of the study. (incl vitamin C, Acetylcysteine)
* Female subjects will take a urinary pregnancy test before each exposure and will be excluded if this is positive.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Vascular vasomotor and fibrinolytic function | 4-6 hours after exposure
  Forearm venous occlusion plethysmography to measure forearm blood flow during unilateral intrabrachial infusion of endothelial-dependent (bradykinin and acetylcholine) and -independent (sodium nitroprusside and verapamil) vasodilators. Fibrinolytic function assessed by blood sampling after infusion of bradykinin for tissue plasminogen activator and plasminogen activator inhibitor-1.

SECONDARY OUTCOMES:
Respiratory function tests | 6 hours after exposure
  Basic spirometry will be performed at baseline and 6 hours after each exposure
Inflammatory markers | Baseline and up to 24 hours after exposure
  Blood samples will be taken and stored as plasma and serum for measurement of inflammatory mediators
Central arterial stiffness | Baseline and post exposure
  Central arterial stiffness (PWV and PWA) will be measured at baseline and immediately after the exposure

CONTACTS AND LOCATIONS:
Overall Officials: Jenny A Bosson Damewood, MD PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University Hospital, Umeå, Sweden

REFERENCES:
- [Derived] Unosson J, Kabele M, Boman C, Nystrom R, Sadiktsis I, Westerholm R, Mudway IS, Purdie E, Raftis J, Miller MR, Mills NL, Newby DE, Blomberg A, Sandstrom T, Bosson JA. Acute cardiovascular effects of controlled exposure to dilute Petrodiesel and biodiesel exhaust in healthy volunteers: a crossover study. Part Fibre Toxicol. 2021 Jun 14;18(1):22. doi: 10.1186/s12989-021-00412-3. PMID 34127003